CLINICAL TRIAL: NCT07126041
Title: End-to-end Digital Transformation for Primary Health Care Performance Management Via Scalable Public Health Empowerment, Research, and Education Sites: A Stepped-Wedge Cluster Randomized Trial
Brief Title: Scalable Public Health Empowerment, Research, and Education Sites (SPHERES)
Acronym: SPHERES
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oxford University Clinical Research Unit Indonesia (Other)
Collaborators: Summit Institute for Development, Indonesia (Other)
Responsible Party: Principal Investigator, Anuraj Shankar, D. Sc., Oxford University Clinical Research Unit Indonesia
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: OUCRU-ID.2025.002; Grant Number : INV-070822 (Other: Gates Foundation funding identifier)
Record Dates: First submitted 2025-08-04; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Pregnancy; Neonatal Mortality; Tuberculosis; Hepatitis B; Hypertension; Diabetes Mellitus
Keywords: Primary health care performance; Digital health transformation; Maternal health; Child health; Immunization; Stunting; Tuberculosis; Hepatitis B; Diabetes mellitus; Hypertension; Health system strengthening; Indonesia; Health governance; Human resource management; Work culture
MeSH Terms: conditions — Tuberculosis; Hepatitis B; Hypertension; Diabetes Mellitus; Growth Disorders | interventions — Prescriptions

STUDY DESIGN:
Intervention Model Description: The study follows a stepped-wedge cluster randomized design in which primary health centers (PHCs) are randomized to receive the intervention in phased steps over time/sequentially. Each cohort enters a digital readiness of up to two months before transitioning into the full SPHERES intervention. Transitions to a new sets of clusters would occur approximately every four months, with full coverage expected within sixteen months of study start.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPHERES Intervention Arm (Experimental): Participants (district populations) receive services improved by the SPHERES model, which includes structured prescription-for-action protocols targeting three priority domains (infectious disease, maternal & child health, and non-communicable diseases).
  Interventions: Other: Prescription for Action (SPHERES Model)
- Control (No Intervention): Standard of care are expected at primary health centers before the SPHERES intervention is deployed

INTERVENTIONS:
Other: Prescription for Action (SPHERES Model) — A system-level intervention consisting of:
  * a digital dashboard displaying local health services, outcome indicators, and operational data in a secure Public Health Data Theater;
  * structured monthly prescription guides targeting service improvements across three priority program areas;
  * monthly performance monitoring with district health leaders. The intervention is applied at the PHC level, all supported by digital capacity building, district-level deployment of implementation teams, and intersectoral secure health data exchange.
  Arms: SPHERES Intervention Arm

SUMMARY:
SPHERES is a health service research trial in the Indonesian primary care system designed to improve health system performance using a structured data-driven action model. The intervention empowers district health leaders to make data-informed decisions that will enhance outcomes across maternal, child, infectious, and non-communicable disease programs.

DETAILED DESCRIPTION:
The SPHERES (Scalable Public Health Empowerment, Research and Education Sites) study is a stepped-wedge health service research trial designed to assess the impact of a complex intervention to enhance the performance of Indonesia's primary health care system through an integrated package of digital health tools to enhance data interoperability, human resource and performance improvement, data-driven decision-making, and changes in work culture toward information-based decision-making, actions, and accountability. The central innovation lies in the "prescription for action" approach, wherein district health managers and heads of primary healthcare centers (PHC) create structured monthly prescriptions that describe actions to be taken to improve primary health care informed by real-time health data visualized on interactive dashboards. These prescriptions are tailored to address gap in priority service delivery challenges including gaps in preventive and promotive care - such as low coverage or quality of antenatal, intrapartum, or postnatal care, or missed opportunities for hepatitis B prevention in pregnancy, or gaps in overall diagnosis and treatment of tuberculosis, or gaps in overall screening and diagnosis and treatment of hypertension or diabetes, - and are grounded in both epidemiological insight and health systems analysis.

As a cluster-randomized stepped-wedge health service trial in the Indonesian primary care system, SPHERES involve multiple primary healthcare centers (PHCs) as the unit of intervention across two districts: West Lombok (West Nusa Tenggara Province) and Purbalingga (Central Java Province). At regular intervals (approximately every 4 months), new clusters (approximately 25% of the total number of PHCs in the district) are transitioned from control to intervention status, until all sites receive the SPHERES intervention within 16 months. This phased approach allows for rigorous evaluation while ensuring equitable access to the program. The intervention package includes: (1) establishment of Public Health Data Theaters as training centers for the active use of data for decision-making using interactive dynamic dashboards, public health data rounds, prescriptions for action for precision public health, digital report cards, and team-based care, (2) deployment of Sustainable Scaling Teams to engage districts in developing the essential technical and management skills for digital ecosystems, and (3) establish ecosystems of interoperable data at the district level to support curative, preventive, and promotive care delivery by frontline health workers. Thus, the intervention will be implemented over 16 months, with approximately 25% of PHCs transitioning every quarter from control to intervention in monthly waves, starting August 2025, with all PHCs receiving the intervention by August 2026.

To support high-fidelity implementation, at each phase of the stepped-wedge, each cluster undergoes a two-phase transformation, a pre-intervention digital readiness phase, followed by the intervention interventions, i.e. the "prescriptions for action" phase. The preparatory step focuses on strengthening digital infrastructure and practices at the PHC level, including standardizing electronic health record inputs, and ensuring interoperability across digital health platforms. Sequencing this digitalization phase ahead of the "prescriptions for action" phase enhances the fidelity and compliance for managerial and behavioral actions that may be included within the "prescriptions for action" intervention.

SPHERES targets improvements in coverage, quality, and outcomes across three priority domains: maternal and child health (including immunization and stunting), infectious disease (tuberculosis and hepatitis B), and non-communicable diseases (diabetes and hypertension). The study will assess impacts on service uptake (e.g., ANC 6 coverage, quality of care, diabetes screening), clinical outcomes (e.g., neonatal mortality, TB treatment success, Hepatitis B vertical transmission), and system-level indicators (e.g., prescription compliance, data use in decision-making). Embedded within the project is a robust capacity-building component for health workers and program managers, along with qualitative assessments of acceptability, feasibility, and perceived value.

SPHERES is expected to produce evidence for improving PHC service quality and responsiveness across Indonesia. By combining routine data analytics with a structured decision-support mechanism, the intervention aims to institutionalize active data use at the district level. Findings from SPHERES are expected to inform Indonesia's Ministry of Health Digital Roadmap and broader digital health transformation strategy and offer generalizable insights into how data empowerment combined with human resource management and change in work culture can drive system-wide improvements in low- and middle-income countries.

ELIGIBILITY:
Inclusion Criteria:

* Residing in or participating in the district catchment areas
* Receiving services from participating health care facilities
* Health providers and district health officials consent to participate in data collection

Exclusion Criteria:

* Individuals (health workers or patients) who decline to provide informed consent.
* Individuals who are not directly involved in or accessing services from health care facilities or district health offices.
* Inability to provide consent due to cognitive impairment or acute illness for health workers or district health officials involved in data collection

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1750000 (Estimated)
Dates: Start 2025-08-14 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Difference in neonatal mortality rate between intervention and control periods | Baseline up to 16 months, with data collected monthly at each site (i.e. baseline, at the end of month 1, at the end of month 2, and so on until at the end of month 16)
  Neonatal mortality per 1,000 live births, calculated using health facility and civil registration data, and community household sampling surveys

SECONDARY OUTCOMES:
Difference in complete antenatal care (ANC 6) visit coverage between intervention and control periods | Baseline up to 16 months, with data collected monthly at each site (i.e. baseline, at the end of month 1, at the end of month 2, and so on until at the end of month 16)
  Percentage of pregnant women completing ≥6 ANC visits calculated using health facility data, paper based registry, and/or community household sampling surveys
Difference in complete basic childhood immunization coverage between the intervention and control period | Baseline up to 16 months, with data collected monthly at each site (i.e. baseline, at the end of month 1, at the end of month 2, and so on until at the end of month 16)
  Proportion of children aged 12-23 months receiving all recommended basic childhood vaccines according to Indonesian Pediatric Society guidelines using health facility data, paper based registry, and/or community household sampling surveys
Difference in TB treatment success rate between intervention and control periods | Baseline up to 16 months, with data collected monthly at each site (i.e. baseline, at the end of month 1, at the end of month 2, and so on until at the end of month 16)
  Percentage of new bacteriologically confirmed TB patients with documented treatment success (cure or completion) calculated using health facility data
Difference in screening coverage for diabetes mellitus among adults between the intervention and control periods | Baseline up to 16 months, with data collected monthly at each site (i.e. baseline, at the end of month 1, at the end of month 2, and so on until at the end of month 16)
  Proportion of adults aged ≥40 screened for random blood glucose or fasting blood glucose calculated using health facility data
Difference in the rate of vertical transmission of hepatitis B between intervention and control periods | Baseline up to 16 months, with data collected monthly at each site (i.e. baseline, at the end of month 1, at the end of month 2, and so on until at the end of month 16)
  Proportion of infants born to hepatitis B surface antigen (HBsAg)-positive mothers who test positive for HBsAg at 9 to 12 months of age. Data will be collected to evaluate the effectiveness of Tenofovir initiation, timely birth dose, routine childhood Hepatitis B vaccination, and HBIG administration as part of the vertical transmission prevention protocol.
Difference in the uptake of dashboard use among district health managers and heads of PHC | Baseline up to 16 months, with data collected monthly at each site (i.e. baseline, at the end of month 1, at the end of month 2, and so on until at the end of month 16)
  Proportion of monthly coordination meetings in which district health managers and heads of PHC accessed and used the SPHERES digital dashboard to review performance data and guide decision-making. Usage will be measured through system access logs and meeting documentation.
Difference in prescription-for-action implementation rate at the PHC | Baseline up to 16 months, with data collected monthly at each site (i.e. baseline, at the end of month 1, at the end of month 2, and so on until at the end of month 16)
  Proportion of prescriptions-for-action issued during Public Health Data Theater sessions that are completed by PHCs within one month. Data will be collected from district monitoring reports and PHC-level follow-up documentation.

CONTACTS AND LOCATIONS:
Overall Officials: Anuraj H Shankar, D. Sc., Principal Investigator — Oxford University Clinical Research Unit Indonesia
Locations (2):
- Indonesia (2):
  - Purbalingga District Health Office, Purbalingga, Central Java
  - West Lombok District Health Office, Gerung, West Nusa Tenggara

IPD SHARING:
Plan to Share IPD: No
The study will not share individual participant data due to the population-level nature of the intervention and national data privacy regulations. Only aggregated and de-identified/anonymized data and codebook may be made publicly available upon publication.
  All data collection, storage, and analysis procedures will comply with Indonesia's Personal Data Protection Law (UU PDP), Ministry of Health guidance, and institutional ethical standards.

REFERENCES:
- See also: Official project website for SPHERES, providing information on project background, implementation framework, partnerships, project status, and the investigators involved. — https://www.oucru.org/project/spheres/